CLINICAL TRIAL: NCT04205838
Title: IL-1 Receptor Antagonist to Prevent Severe Chimeric Antigen Receptor T-Cell Related Encephalopathy Syndrome
Brief Title: Anakinra in Preventing Severe Chimeric Antigen Receptor T-Cell Related Encephalopathy Syndrome in Patients With Recurrent or Refractory Large B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-000604; NCI-2019-02887 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-000604 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2019-10-02; First posted 2019-12-20 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma; Progressive Disease; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Recurrent Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Refractory Transformed Follicular Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Disease Progression | interventions — Interleukin 1 Receptor Antagonist Protein; Receptors, Interleukin-6; axicabtagene ciloleucel; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Prevention (anakinra, CAR T-cell therapy) (Experimental): Patients receive standard lymphodepleting therapy including fludarabine and cyclophosphamide on days -5 to -3, then receive axicabtagene ciloleucel CAR T-cell infusion. Patients with clinical evidence of ICANS of any grade, or CRS >= grade 3 receive anakinra SC every 6-12 hours for 12-36 doses over 9 days in the absence of unacceptable toxicity.
  Interventions: Biological: Anakinra; Biological: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate

INTERVENTIONS:
Biological: Anakinra — Given SC
  Other Names: Kinaret; Kineret; rIL-1ra; rIL1RN
Biological: Axicabtagene Ciloleucel — Given via infusion
  Other Names: KTE C19; KTE-C19; KTE-C19 CAR; Yescarta
Drug: Cyclophosphamide — Given via infusion
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given via infusion
  Other Names: Fluradosa
Drug: Fludarabine Phosphate — Given via infusion
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586

SUMMARY:
This phase II trial studies how well anakinra works in preventing severe chimeric antigen receptor T-cell-related encephalopathy syndrome after chimeric antigen receptor T-cell therapy in patients with large B-cell lymphoma that has come back or has not responded to treatment. Immunosuppressive therapy, such as anakinra, is used to decrease the body?s immune response, which may prevent severe chimeric antigen receptor T-cell-related encephalopathy syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if it is feasible to accrue a sufficient number of study participants at one site, in order to justify expanding the trial to three additional sites (pilot study).

II. To estimate the efficacy of anakinra in prevention of severe immune effector cell-associated neurotoxicity syndrome. syndrome (ICANS) (full study).

SECONDARY OBJECTIVES:

I. To estimate the impact that anakinra has on the efficacy of chimeric antigen receptor (CAR) T-cell therapy for relapsed/refractory lymphoma.

II. To estimate the rate of subsequent ICANS development in patients who receive anakinra for grade >= 3 cytokine release syndrome (CRS) in the absence of ICANS.

III. To estimate the duration of neurotoxicity in patients who receive anakinra.

IV. To estimate the duration of severe neurotoxicity in patients who receive anakinra.

V. To determine if anakinra causes persistent hepatotoxicity in patients receiving CAR T-cell for refractory lymphoma.

VI. to evaluate the overall toxicity of anakinra in patients receiving CAR T-cell therapy for refractory lymphoma.

EXPLORATORY OBJECTIVES:

I. To evaluate CRS and ICANS grade by using the American Society for Blood and Marrow Transplantation (ASBMT) 2018 consensus grading for adults.

II. To investigate changes in inflammatory markers including IL-1 and IL-6 in the peripheral blood during episodes of ICANS.

III. To describe the electroencephalogram (EEG) changes that characterize ICANS.

OUTLINE:

Patients receive standard lymphodepleting therapy including fludarabine and cyclophosphamide on days -5 to -3, then receive axicabtagene ciloleucel CAR T-cell infusion. Patients with clinical evidence of ICANS of any grade, or CRS >= grade 3 receive anakinra subcutaneously (SC) every 6-12 hours for 12-36 doses over 9 days in the absence of unacceptable toxicity.

After completion of study, patients are followed up at 30, 90, and 100 days, then at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory large B-cell lymphoma that has progressed on two prior lines of therapy, who meet the indication for the Food and Drug Administration (FDA)-approved therapy axicabtagene ciloleucel
* Large B-cell lymphoma includes diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, and DLBCL arising from follicular lymphoma
* The above includes patients with progressive or stable disease as the best response to the most recent treatment regimen or disease progression within 12 months after autologous hematopoietic stem cell transplantation
* Patients with central nervous system (CNS) involvement of large B-cell lymphoma that originated outside of the CNS will be included (not primary CNS lymphoma)
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) =< 2.5 upper limit of normal
* Total bilirubin =< 2.0 mg/dL
* Creatinine clearance > 30 mL/min based on Cockcroft-Gault formula
* Patients with human immunodeficiency virus (HIV) who have an undetectable viral load will be included
* Deemed competent to make medical decisions

Exclusion Criteria:

* Patients who receive CAR T-cell therapy with a product other than axicabtagene ciloleucel
* Primary CNS lymphoma
* Transformed DLBCL from chronic lymphocytic leukemia (CLL)
* Burkitt?s lymphoma
* Bridging chemotherapy completed < 7 days prior to CAR T-cell lymphodepleting chemotherapy
* In patients who receive bridging chemotherapy, positron emission tomography (PET)-computed tomography (CT) or CT of chest, abdomen, pelvis was not done after bridging chemotherapy prior lympho-depleting therapy
* Most recent PET-CT or CT of all known disease is sites done more than 6 weeks prior to CAR T-cell infusion
* Any individual CNS tumor mass > 2 cm
* History of autologous hematopoietic stem cell transplantation administered less than 100 days prior to CAR T-cell infusion
* History of allogeneic hematopoietic stem cell transplantation
* Treatment with alemtuzumab within 6 months prior to leukapheresis, or treatment with clofarabine or cladribine within 3 months prior to leukapheresis
* Less than 3 half-lives elapsed since receiving immune checkpoint inhibitor (pembrolizumab, ipilimumab, nivolumab, atezolizumab, etc.)
* Presence of uncontrolled fungal, bacterial, or viral infection that require intravenous (IV) antimicrobial treatment
* History of autoimmune disease resulting in end-organ damage, or autoimmune disease requiring systemic immunosuppressants or disease-modifying antirheumatic drug (DMARDs) within the past 6 months
* Hypersensitivity to E. Coli-derived proteins
* Patients with HIV who have a detectable viral load
* Pregnant or nursing
* Fertile women who decline use of contraception during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients who met the eligibility criteria to receive and did receive anakinra | Up to 12 months
  The study will be considered feasible if 8 study participants are enrolled over 12 months at University of California, Los Angeles.
Rate of severe chimeric antigen receptor T-cell-related encephalopathy syndrome (ICANS) | Up to 30 days
  Will be defined as grade >= 3 neurotoxicity by Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03. The proportion of patients developing severe ICANS and the corresponding 90% binomial exact confidence interval (CI) will be reported.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 90 days
  Will be defined as a complete response or partial response per the International Working Group criteria malignancy lymphoma based on positron emission tomography (PET)/computed tomography (CT) scan. To account for the adaptive nature of Simon?s two-stage design, final analysis of the objective response rate will report the uniformly minimum variance unbiased estimator and the corresponding p-value and 95% CI for the ORR.
Proportion of patients who received anakinra and develop ICAN | Up to 30 days
  The proportion of patients who received anakinra in the absence of ICANS and then develop ICANS of any grade out of the total number of participants who received anakinra in the absence of ICANS will be evaluated. Will be summarized using descriptive statistics such as proportion, mean, standard deviation, median, as appropriate.
Duration of neurotoxicity | From first day of CRES of any grade to complete resolution of CRES, assessed up to 100 days
  Defined as number of days that elapse from first day of ICANS of any grade to complete resolution of ICANS. Will be summarized using descriptive statistics such as proportion, mean, standard deviation, median, as appropriate.
Duration of neurotoxicity | From first day of ICANS of >= grade 3 to improvement of ICANS to < grade 3, assessed up to 100 days
  Defined as number of days that elapse from first day of ICANS of >= grade 3 to improvement of ICANS to < grade 3 based on CTCAE v4.03. Will be summarized using descriptive statistics such as proportion, mean, standard deviation, median, as appropriate.
Persistent hepatotoxicity | Up to 100 days
  Will be defined as grade > 2 aspartate aminotransferase (AST)/alanine aminotransferase (ALT) increased for at least 4 weeks duration according to CTCAE v4.03. Will be summarized using descriptive statistics such as proportion, mean, standard deviation, median, as appropriate.
Incidence of adverse events (AEs) | Up to 100 days
  Will be based on CTCAE v4.03. Will be summarized using descriptive statistics such as proportion, mean, standard deviation, median, as appropriate. All AEs will be listed, documenting the course, outcome, severity, and relationship to the study treatment. Incidence rates of AEs and the proportion of subjects prematurely withdrawn from the study due to AEs will be shown.

OTHER OUTCOMES:
ICANS grade | up to 30 days
  Will evaluate ICANS grade by using the American Society for Blood and Marrow Transplantation 2018 consensus grading for adults.
Cytokine release syndrome (CRS) grade | Up to 30 days
  Will evaluate CRS grade by using the American Society for Blood and Marrow Transplantation 2018 consensus grading for adults.
Changes in inflammatory markers | Baseline up to 6 days following initiation of anakinra
  Peak median serum blood and cerebral spinal fluid (CSF) levels of IL-1 and IL-6 will be summarized using descriptive statistics or contingency tables, as appropriate.
Changes in Electroencephalogram (EEG) that characterize ICANS: Slowing of EEG activity. | Baseline up to 100 days
  Slowing of EEG activity including waveform, spectrum, spectrogram, and power in the slow (0.1-1 Hz), delta (1 to 4 Hz), theta (4 to 8 Hz) bands.
Changes in Electroencephalogram (EEG) that characterize ICANS: focal slowing | Baseline up to 100 days
  Changes in Electroencephalogram (EEG) that characterize ICANS: Focal regional slowing of the EEG activity within the frontal, temporal, parietal, or occipital region in the delta (<4Hz) and/ or theta (4-8 Hz) band.
Changes in Electroencephalogram (EEG) that characterize ICANS: periodic discharge | Baseline up to 100 days
  Generalized or lateralized or bilateral independent or multifocal periodic discharges (repetitive discharges with similar morphology and recurring at regular or near-regular inter-discharge intervals)
Changes in Electroencephalogram (EEG) that characterize ICANS: rhythmic activity | Baseline up to 100 days
  Generalized or lateralized or bilateral independent or multifocal Rhythmic delta activity (</= 4 Hz).
Changes in Electroencephalogram (EEG) that characterize ICANS: Generalized or lateralized or bilateral independent or multifocal spike | Baseline up to 100 days
  Generalized or lateralized or bilateral independent or multifocal spike (duration of the wave <70ms) or sharp (duration of the wave 70-200ms) discharges.
Changes in Electroencephalogram (EEG) that characterize ICANS: seizures | Baseline up to 100 days
  Electrographic seizure occurrence: Percentage of subjects who experience electrographic seizure while undergoing continuous-EEG monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: John M Timmerman, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - UC Davis Comprehensive Cancer Center, Davis, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California